CLINICAL TRIAL: NCT05603949
Title: Development of Three-dimensional Deep Learning for Automatic Design of Skull Implants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Yau-Zen Chang, Professor, Chang Gung Memorial Hospital
Other Study IDs: 202201082B0
Record Dates: First submitted 2022-09-07; First posted 2022-11-03 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Skull Defect
Keywords: Deep Neural Networks;3D Shape Inpainting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- experimental group
  Interventions: Device: 3D deep learning neural network system

INTERVENTIONS:
Device: 3D deep learning neural network system — With the consent of the patient, we will assist in the production of images of 3D defect blocks for free (3D deep learning neural network system (3D DNN) system process planning), complete the repair and reconstruction under the clinical routine surgery, and track the repair results after surgery. meet medical needs.

SUMMARY:
This project aims to develop an effective deep learning system to generate numerical implant geometry based on 3D defective skull models from CT scans. This technique is beneficial for the design of implants to repair skull defects above the Frankfort horizontal plane.

DETAILED DESCRIPTION:
Designing a personalized implant to restore the protective and aesthetic functions of the patient's skull is challenging. The skull defects may be caused by trauma, congenital malformation, infection, and iatrogenic treatments such as decompressive craniectomy, plastic surgery, and tumor resection. The project aims to develop a deep learning system with 3D shape reconstruction capabilities. The system will meet the requirement of designing high-resolution 3D implant numerical models efficiently.

A collection of skull images were used for training the deep learning system. Defective models in the datasets were created by numerically masking areas of intact 3D skull models. The final implant design should be verified by neurosurgeons using 3D printed models.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for cranioplasty
2. Informed consent

Exclusion Criteria:

(1)No informed consent

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Take a medical center as the research object
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Number of patients where there is no need to adapt the Patient Specific Implant (PSI) edges | 6 weeks after surgery by standardised questionnaire
  Number of patients where there is no need to adapt the Patient Specific Implant (PSI) edges
Number of patients where there is no need to augment/fill clefts between the Patient Specific Implant (PSI) and patient´s bone | 6 weeks after surgery by standardised questionnaire
  Number of patients where there is no need to augment/fill clefts between the Patient Specific Implant (PSI) and patient´s bone

CONTACTS AND LOCATIONS:
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taoyuan, Taiwan